CLINICAL TRIAL: NCT06200610
Title: Study of Prevalence of the Covid-19 Among the Staff of the Emergency Department
Acronym: ED-Covid-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8018
Record Dates: First submitted 2023-12-22; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: Covid-19; COVID-19 Pandemic; Emergency services
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since December 2019, a new coronavirus, SARS-CoV-2, has been identified in the city of Wuhan in Hubei province in China and is the cause of a global pandemic. This highly contagious virus is responsible for the COVID-19 disease, the manifestations of which can range from a simple flu-like syndrome to acute respiratory distress syndrome (ARDS). Transmission of SARS-CoV-2 is mainly linked to droplets. The mode of transmission of SARS-CoV-2 involves at least droplet-type isolation for caregivers with wearing a surgical mask and extended contact type (overcoats, caps, gloves). During procedures with a high risk of aerosolization of viral particles (intubation, aerosols, aspirations, nasopharyngeal swabs), wearing an FFP2 mask and protective glasses are recommended. In addition, oxygen therapy, particularly at a flow rate greater than 6 L/min, could also lead to airborne contamination.

The occupational risk of contamination of health professionals is well identified, particularly in Chinese but also Italian studies. In Italy, 20% of healthcare workers have been contaminated. In China, a rate of 3.5 to 29% in Wuhan hospitals has been identified.

Among the professionals exposed within the hospital, those in emergency services are part of the category with the greatest risk of contamination along with those in intensive care units. Recommendations from experts from the French intensive care society and foreign companies made it possible to identify the situations most at risk of contamination. In addition, the organization has made it possible to better understand patient care circuits in order to limit the risks of contamination. However, procedural errors may exist, implying the need for frequent training sessions for professionals. In addition, if the recommendations specify the need to obtain negative pressure in the rooms or at least zero, the material limits linked to reception in emergency departments with the need for intubation of a significant number of patients sometimes makes it difficult to carry out these risky actions under optimal conditions. Finally, the methods of sorting suspected cases to organize care in areas different from other emergency patients do not prevent assignment errors, a source of contamination for caregivers and patients.

Thus, health professionals are among the priority people to be screened in accordance with the recommendations of the High Authority of Health. Indeed, even if symptomatic healthcare workers were mostly screened at least by taking a nasopharyngeal swab, some healthcare workers were able to develop immunity to the disease without having been symptomatic. The number of asymptomatic cases of COVID-19 is significant, but the proportion is not yet clearly identified. In addition, massive screening of symptomatic and non-symptomatic healthcare workers would make it possible to reduce the number of nososcomial contamination. Determining the serological status of healthcare workers is a priority, particularly in services on the front line of caring for patients with COVID-19, such as emergency structures.

DETAILED DESCRIPTION:
The aim of the study is to study the seroprevalence of SARS-CoV2 among healthcare personnel in the emergency services of the Strasbourg University Hospitals and the Besançon University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old)
* Part of the emergency staff of the HUS or Besançon University Hospital having worked during the period of the covid-19 pandemic, from March 1, 2020 to May 31, 2020.
* Having carried out serology within the framework of the recommendations of the High Authority of Health of May 2, 2020 on the screening of caregivers
* Having given consent for its biological resources to be reused for research purposes

Exclusion Criteria:

* Subject having expressed opposition to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years old) part of the emergency staff of the HUS or Besançon University Hospital having worked during the period of the covid-19 pandemic, from March 1, 2020 to May 31, 2020, and Having carried out serology within the framework of the recommendations of the High Authority of Health of May 2, 2020 on the screening of caregivers
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Presence of antibodies specific to SARS-CoV2 in the serum in the subjects studied | Through study completion, an average of 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Accueil des Urgences - CHU de Strasbourg - France, Strasbourg, France